CLINICAL TRIAL: NCT07138261
Title: Taiwanese Anaplastic Thyroid Cancer Registry
Acronym: TATC
Status: Not yet recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: T1325
Record Dates: First submitted 2025-08-03; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Carcinoma, Anaplastic
Keywords: Anaplastic thyroid cancer; Genetic aberrations in anaplastic thyroid cancer; Treatment for anaplastic thyroid cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The archived tumor sample of FFPE blocks derived from biopsy or surgery is applied from each hospital. For each tumor sample, 10 slices of 4um are needed with 3 put in non-coated slides and 7 in coated slides. Another 10 slides of 4um of non-coated slides will be collected for NGS-based study if there is other funding support available.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- anaplastic thyroid cancer (ATC): Pathologically or cytologically confirmed ATC and diagnosed after 2015.

SUMMARY:
Primary treatment strategies for ATC have included surgical resection combined with radiotherapy, chemotherapy, or concurrent chemoradiation therapy. Despite these aggressive approaches, disease recurrence or progression remains frequently observed. Recent advances in molecular diagnostics and targeted therapy development have expanded treatment options for ATC patients with actionable genetic alterations, such as BRAF mutations or NTRK fusions. Nevertheless, for patients lacking identifiable targetable mutations, therapeutic options remain limited and clinical outcomes are poor. To address this unmet clinical need, the investigators aim to analyze baseline characteristics, treatment outcomes, and biomarker profiles from a larger cohort of ATC patients, with the goal of identification of predictive biomarkers and potential therapeutic targets. Given the rarity of ATC, conducting comprehensive studies at a single institution is challenging. Therefore, the investigators propose to establish a multi-center registry to systematically collect clinical data and tumor specimens from ATC patients.

DETAILED DESCRIPTION:
Thyroid cancers are pathologically classified into differentiated thyroid cancer (DTC),medullary (MTC) and anaplastic carcinoma (ATC). ATC accounts for approximately 1% of thyroid cancer cases in Taiwan and is characterized by its aggressive clinical course with extremely poor prognosis. A subset of patients may present with mixed histology, exhibiting both DTC and ATC components, or may experience progression from DTC to ATC. These cases are typically associated with rapid disease progression and significantly worse clinical outcomes. Because the incidence of ATC is very low, it is not easy to conduct clinical trials with large sample size to investigate novel treatment strategies with some effective treatment modalities reported by case reports or case series. Recently, the genetic test has been reimbursed by our health Bureau for ATC cases. In this study, the investigators aim to enroll ATC patients from multi-centers in Taiwan to collect the baseline characteristics, genetic data, treatment patterns, and clinical outcome of the ATC patients. In addition, the investigators want to collect tumor and blood samples for ATC patients to explore the biomarkers and potential treatment modalities from the real-world data.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed ATC and diagnosed after 2015.
2. Capable of understanding and complying with the protocol requirements and signed informed consent. The dead patient can be enrolled without signed informed consent and they were dead before 2025.6.30.

Exclusion Criteria:

1. Inability and unwillingness to give informed consent except dead patient.
2. Patients refuse for collection of clinical data and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were pathologically or histologically diagnosed as anaplastic thyroid cancer (ATC) are the target population. The ATC may be transformed from DTC or de novo cases. Anticipated 100 patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2035-12-30 (Estimated); Study Completion 2035-12-30 (Estimated)

PRIMARY OUTCOMES:
Enrolled more than 100 anaplastic thyroid cancer patients | Pathologically or cytologically confirmed ATC and diagnosed after 2015，The dead patient can be enrolled without signed informed consent and they were dead before 2025.6.30.
  100 anaplastic thyroid cancer patients, including denovo ATC or ATC transformed from DTC, or co-existence of ATC and DTC.

SECONDARY OUTCOMES:
To reported of survival with demographic characteristics, treatment patterns and tumor and blood samples for further biomarker of ATC in Taiwan. | After registration. The clinical data of treatment, treatment response, treatment toxicities, and survival of the enrolled patients after enrollment will be collected every 3 months. Followed up for the survival till 3 years.
  Patients with histologically or cytologically diagnosed anaplastic thyroid cancer are eligible. Eligible patients will be enrolled to collect the clinical data,genetic data, treatment and outcomes of the patients, and blood and archived tumor samples. The clinical data include baseline characteristics, diagnosis,stage, prior and current treatment, and treatment outcome (response, toxicities and survival). The genetic data includes any genetic data performed by IHC,sanger sequencing or NGS-based oncopanel or other approaches. The archived tumor sample will be collected for further biomarker study. A blood sample will also be collected for germline mutation analysis. The clinical and genetic data collected in this trial will be stored in the Clinical Trial Information Management System (CTIMeS) of Taiwan Cooperative Oncology Group (TCOG) for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu Taiwan Cooperative Oncology Group,NHRI,Taipei, Taiwan, M.D. PhD, Study Chair — Taiwan Cooperative Oncology Group,NHRI,Taipei, Taiwan; Hui-Jen Tsai Taiwan Cooperative Oncology Group,NHRI,Taipei, Taiwan, M.D. PhD, Principal Investigator — Taiwan Cooperative Oncology Group,NHRI,Taipei, Taiwan
Locations (9):
- Taiwan (9):
  - Taipei Veterans General Hospital, Taipei, Taiwan/Taipei
  - Kaohsiung Medical University, Kaohsiung City
  - National Taiwan University Hospital ,NTUH Hsin-Chu Branch, Sindian City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - CHANG GUNG MEMORIAL HOSPITAL, Linkou, Taoyuan District

REFERENCES:
- [Background] Smallridge RC, Ain KB, Asa SL, Bible KC, Brierley JD, Burman KD, Kebebew E, Lee NY, Nikiforov YE, Rosenthal MS, Shah MH, Shaha AR, Tuttle RM; American Thyroid Association Anaplastic Thyroid Cancer Guidelines Taskforce. American Thyroid Association guidelines for management of patients with anaplastic thyroid cancer. Thyroid. 2012 Nov;22(11):1104-39. doi: 10.1089/thy.2012.0302. PMID 23130564
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- See also: Cancer Registry Annual Report, 2022 Taiwan. Health Promotion Administration Ministry of Health and Welfare — https://www.hpa.gov.tw/EngPages/Detail.aspx?nodeid=1070&pid=16384